CLINICAL TRIAL: NCT04398823
Title: A Multicenter Prospective Clinical Study of Endoscopic Foam Sclerotherapy for Internal Hemorrhoids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Tongren Hospital,Shanghai Jiao Tong University School of Medicine (Unknown); Shanghai Construction Group Hospital (Unknown); Shandong Maternal and Chidl Care Service Center (Unknown); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); West China Fourth Hospital, Sichuan University (Unknown); The First Hospital of Anhui Medical University (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Jiangsu Provincial Second Chinese Medicine Hospital (Unknown); Anhui Provincial Hospital (Other Government); Luoyang Central Hospital (Other); Ganzhou Fifth pepole's Hospital (Unknown); Changzhi People's Hospital (Other); Nanjing PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH-20-006
Record Dates: First submitted 2020-05-09; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-04

CONDITIONS: Grade/Stage I Hemorrhoids; Prolapsed Grade II Internal Haemorrhoid; Prolapsed Grade III Internal Haemorrhoid
Keywords: hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam sclerotherapy,FS (Active Comparator): Participants in this arm will receive the enteroscopic treatment with the sclerosing foam of lauromacrogol.
  Interventions: Drug: Sclerosing foam of Lauromacrogol
- Liquid sclerotherapy,Ls (Placebo Comparator): Participants in this arm will receive the enteroscopic treatment with the liquid of lauromacrogol.
  Interventions: Drug: Sclersing liqiud of Lauromacrogol

INTERVENTIONS:
Drug: Sclerosing foam of Lauromacrogol — Participants in FS will receive enteroscopy with the sclerosing foam of lauromacrogol.
  Arms: Foam sclerotherapy,FS
Drug: Sclersing liqiud of Lauromacrogol — Participants in LS will receive enteroscopy with the sclerosing liquid of lauromacrogol.
  Arms: Liquid sclerotherapy,Ls

SUMMARY:
"Internal hemorrhoid" affects the quality of life due to hemorrhage and prolapse as a common and frequently-occurring disease. Endoscopic sclerosing agent injection has replaced traditional surgery and become the most commonly used treatment method in developed countries. At present, how to reduce the side effects of sclerosing agent and accurately determine the injection site and depth has become a difficult clinical problem. The research group creatively put forward the theory of foam sclerosing agent to treat internal hemorrhoids in the early stage. With the aid of transparent cap, the visibility of surgical field of vision can be improved. The mini probe ultrasound (MPS) is proposed to effectively evaluate the submucosal in

ELIGIBILITY:
Inclusion Criteria:

* People are willing to sign the informed consent form of this trial.
* People(aged 18 to 70 years) with clinical symptoms such as bleedingprolapse and so on have been diagnosed with grade I, grade II and grade III internal hemorrhoids by colonic epdoscopy;
* People can follow short-term (3 month) and long-term (12 month) visit plans;
* Describe symptoms objectively and actively complete the evaluation scale;
* No allergic diseases and allergy to sclerosing drugs;
* Non-lactating and pregnant women: patients without pregnancy plan (including the men) in 1 month after the test;
* Did not participate in any drug trials (including this trial drug) within 3 months before the trial;
* People with long-term use of anticoagulant drugs (such as aspirin, clopidogrel, etc.) need to be stopped for 5-7 day

Exclusion Criteria:

* People with severe insufficiency of heart, brain, lung and other organs, leading to inability to tolerate endoscopic treatment;
* People with drug allergies or abnormal blood coagulation function;
* People suffering from or combined with digestive tract diseases,such as the colon malignancyulcerative colitis or Crohn's diseaseacute diarrheaacute thrombotic internal hemorrhoids with painanal fistulaanal fissurefecal incontinence
* Men with history of severe prostate hypertrop;
* People with any reasons that the researchers believe can not be selected

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the condition of bleeding、perianal pruritus 、the degree of prolapse of internal hemorrhoids and the influence of internal hemorrhoids by self-assessment. | 12 months
  After 12 months,all the participants will receive the telephone follow-up to record their self-assessment.
the condition of perianal pruritus、the description of hemorrhoids(include the number and depth of hemorrhoids)、the need for additiongal sclerotherapy under colonic endoscopy. | 12 months
  after 12 months ,all the participants will receive the colonic endoscopy and we will record the degree of prolapse of internal hemorrhoids、the numbers of hemorrhoid under colonic endoscopy.

SECONDARY OUTCOMES:
the condition of participants' bleeding、perianal pain and perianal pruritus after the endoscopic treatment. | 1 day
  one day after receiving endoscopic treatment , all the participants will receive the telephone follow-up and we will record their self-assessment,include the condition of bleeding、perianal pain and perianal pruritus.
the condition of bleeding、perianal pruritus 、the degree of prolapse of internal hemorrhoids and the influence of internal hemorrhoids by self-assessment. | 3 months
  After 3 months,all the participants will receive the telephone follow-up to record their self-assessment.
the condition of participants' bleeding、perianal pain and perianal pruritus after the endoscopic treatment. | 1 week
  one week after receiving endoscopic treatment , all the participants will receive the telephone follow-up and we will record their self-assessment,include the condition of bleeding、perianal pain and perianal pruritus.
the condition of perianal pruritus、the description of hemorrhoids(include the number and depth of hemorrhoids)、the need for additiongal sclerotherapy under colonic endoscopy. | 3 months
  after 3 months ,all the participants will receive the colonic endoscopy and we will record the degree of prolapse of internal hemorrhoids、the numbers of hemorrhoid under colonic endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Leiming Xu, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Yi Zhang, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Zhenzhong Deng, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Haixia Peng, Principal Investigator — Tong Ren Hospital affiliated to Shanghai Jiaotong University School of Medicine; Hui Pan, Principal Investigator — Shanghai Construction Group Hospital; Fengyu Gao, Principal Investigator — Shandong Maternal and Child Health Center affiliated to Shandong University; Hao Zhang, Principal Investigator — BaoShan People's Hospital
Locations (1):
- Xinhua Hospital,Shangha Jiao Tong University, Shanghai, China